CLINICAL TRIAL: NCT02870270
Title: Prospective Studies on Saliva, Microflora, Diet, Oral Status and Quality of Life in Subjects Undergoing Radiation Therapy in the Head and Neck Region
Brief Title: Prospective Studies on Oral Health and Quality of Life in Head and Neck Cancer Patients
Status: Completed | Type: Observational
Sponsor: Göteborg University (Other)
Collaborators: The Health & Medical Care Committee of the Regional Executive Board, Region Västra Götaland (Unknown)
Responsible Party: Sponsor
Other Study IDs: 682-07
Record Dates: First submitted 2016-08-12; First posted 2016-08-17 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Mouth Diseases; Quality of Life; Secretion; Salivary Gland, Deficient
Keywords: saliva; microflora; diet; quality of life; oral cancer
MeSH Terms: conditions — Mouth Diseases; Mouth Neoplasms | interventions — Antineoplastic Protocols

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Minor salivary gland secretion, stimulated whole saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Head and neck cancer patients: Patients with head and neck cancer who were ≥ 18 years old and had ≥ 16 teeth and no removable prosthesis or dental implants consisting of more than one teeth were included
  Interventions: Other: Cancer treatment

INTERVENTIONS:
Other: Cancer treatment — Patients undergoing treatment for cancer in the head and neck region

SUMMARY:
Radiation therapy (RT) leads to a markedly reduced salivary secretion rate, which makes it difficult to eat and talk and it is a risk factor for oral disorders such as caries and mucosal infections. A reduced salivary secretion rate is often a life long side-effect of the treatment that seriously affect the quality of life. To reduce these side-effects the patients get preventive and supportive oral treatment in connection with their cancer treatment. However, regardless of radiation doses given, the severity of the problems vary considerably. Therefore, a better understanding on when and why problems occur is important for the identification of subjects at risk and to find better measures and treatments, suited for their individual needs.

Dentate subjects were included referred before RT. Data were collected before and during treatment as well as 6, 12 and 24 months after completed RT. Cancer diagnosis, treatment, radiation doses, infections and medication were obtained from medical records.

Dietary habits were registered using a questionnaire focusing on intake of carbohydrate-rich food-items and items containing sugar-substitutes. The subjects weight was registered before, during and after RT.

A clinical examination was performed before and 6, 12 and 24 months after completed RT. Panoramic x-rays were taken as well as bitewing radiographs. The number of teeth, caries status, oral hygiene were registered. Mucositis was registered during RT.

Secretion of stimulated whole saliva was determined. Minor labial and buccal gland saliva secretion rate was determined using the Periotron-method. Microbial samples were collected from the tongue, buccal mucosa and supragingival plaque and microorganisms associated with oral health and oral disorders analysed using cultivation technique.

The quality of life was registered using the questionnaires EORTC QLQ-C30 (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire). To address additional symptoms associated specifically with cancer in the head and neck region and its treatment, a complementary 35-item module, the EORTC QLQ-H&N35 was used.

The patients also completed the Hospital Anxiety and Depression Scales, HADS, which is used to measure severity of anxiety and depressive symptoms and provides estimates of possible mood disorders in patients with somatic comorbidity.

DETAILED DESCRIPTION:
In Europe, about 73 000 persons/year get cancer in the head and neck region. The treatment for oral cancer vary depending on tumour site and stage. Some subjects undergo surgery, some subjects are treated with chemotherapy in combination with the radiation and in some cases brachytherapy is used. Radiation therapy leads to a markedly reduced salivary secretion rate, which makes it difficult to eat and talk and it is a risk factor for oral disorders such as caries and mucosal infections. A reduced salivary secretion rate is often a life long side-effect of the treatment that seriously affect the quality of life. To reduce these side-effects the patients get preventive and supportive oral treatment in connection with their cancer treatment. However, regardless of radiation doses given, the severity of the problems vary considerably. Therefore, a better understanding on when and why problems occur is important for the identification of subjects at risk and to find better measures and treatments, suited for their individual needs.

Dentate subjects referred to Dr. Bodil Fagerberg-Mohlin, before radiation therapy in the head and neck region are included. Data are collected at 5 occasions: before and during treatment as well as 6, 12 and 24 months after completed radiation therapy.

The subjects' cancer diagnosis, treatment, radiation doses, infections and medication are obtained from their medical records. Their odontological preventive treatment and use of other agents with fluoride such as saliva-stimulating chewing gum and tablets are registered.

Dietary habits are registered using a questionnaire focusing on intake of carbohydrate-rich food-items and items containing sugar-substitutes. The subjects are asked to fill in how often they use the items on a 6-grade scale. The subjects weight is registered before, during and after radiation therapy.

A clinical examination is performed before and 6, 12 and 24 months after completed radiation therapy. Panoramic x-rays are taken as well as bitewing radiographs. The number of teeth, caries status, oral hygiene are registered. Mucositis is registered during radiation therapy.

Secretion of stimulated whole saliva is determined before and after radiation therapy. Minor labial and buccal gland saliva secretion rate is determined using the Periotron-method. Centrifuged stimulated saliva and minor gland saliva is stored in the freezer pending analysis of IgA, albumin, mucins and lactoferrin using ELISA-techniques.

Microbial samples are collected at all occasions from the tongue, buccal mucosa and supragingival plaque. The total viable count is registered as well as microorganisms associated with oral health (streptococci, Neisseria), gingival inflammation (Fusobacterium nucleatum, Prevotella), caries (mutans streptococci, lactobacilli) and mucosal infections (Candida, staphylococci, Gram-negative enteric rods and enterococci). The samples are analysed using cultivation technique.

The quality of life is registered using the questionnaires EORTC QLQ-C30 (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire), which is a cancer-specific questionnaire that evaluates health-related quality of life in cancer patients. The questionnaire consists of five function scales, a global quality of life scale, three symptom scales and six single items, in total 30 questions that describe the patients' symptoms and functional level during the prior week. To address additional symptoms associated specifically with cancer in the head and neck region and its treatment, a complementary 35-item module, the EORTC QLQ-H&N35 is used. Both questionnaires have been proved to be reliable and valid. Calculated scale scores range from 0-100. On the functioning scales and Global quality of life scales, a score of 100 represents maximum functioning, whereas on the symptom scales and single items, a score of 100 indicates the worst possible symptoms. For the EORTC questionnaires, a change in score over time >10 can be considered to detect a clinically significant difference.

Hospital Anxiety and Depression scales The patients also complete the Hospital Anxiety and Depression Scales, HADS, which is used to measure severity of anxiety and depressive symptoms and provides estimates of possible mood disorders in patients with somatic comorbidity. HADS is a valid and reliable instrument. The HAD scales consists of 14 items, seven items for depression and 7 items for anxiety with a score range from 0-21. For each factor, the results are interpreted as follows: 8-10 points indicates cases of possible anxiety or depression and >10 points indicates probable anxiety or depression.

Statistical analysis Changes between baseline and 6 months, between 6 and 12 months and between 12 and 24 months will be made using paired samples tests. For analysis of changes within the cancer group, partial correlation will be used analysing associations over time (correlation coefficients of r > 0.4 is considered statistically significant). For quality of life data, a change in score over time of > 10 points could be interpreted as clinically significant. For analysis of associations between QoL and oral status at 6, 12 and 24 months partial correlations will be used (r > 0.4 is considered statistically significant).

ELIGIBILITY:
Inclusion Criteria:

18 years or older

16 or more own teeth

No removable prosthesis

No dental implants consisting of more than one tooth

Able to read and understand Swedish

Exclusion Criteria:

< 18 years old

< 16 teeth

Removable prosthesis

Dental implants consisting of more than one tooth

Severe cognitive impairment

Unable to read and/or understand Swedish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were diagnosed with cancer in the head and neck region and were treated with curative radiotherapy at Sahlgrenska university hospital, Gothenburg, Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2008-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Changes in salivary secretion rate | Pretreatment- two years post treatment

SECONDARY OUTCOMES:
Changes in oral microflora | Pretreatment- two years post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Annica Almståhl, Assoc. prof, Principal Investigator — Göteborg University
Locations (1):
- Institute of odontology, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Almstahl A, Alstad T, Fagerberg-Mohlin B, Carlen A, Finizia C. Explorative study on quality of life in relation to salivary secretion rate in patients with head and neck cancer treated with radiotherapy. Head Neck. 2016 May;38(5):782-91. doi: 10.1002/hed.23964. Epub 2015 Jun 20. PMID 25537660